CLINICAL TRIAL: NCT07178561
Title: The Effect of Physical Activity Program Along With Exercises on Disability Level and Mental Health Among the Elderly Population With Chronic Low Back Pain. Give me Breif Title
Brief Title: Physical Activity and Exercise for Disability and Improving Mental Health in Elderly With Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mosab ALdabbas, Assistant professor at Al azhar university and field officer at ICRC, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Al-Azhar UNIVERSITY in GAZA PA
Record Dates: First submitted 2025-08-27; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; Elderly; sleep; mental health
MeSH Terms: conditions — Psychological Well-Being | interventions — Exercise; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group receive Exercises (Experimental): Exercise and Physical Activity Program for Elderly with Chronic Low Back Pain
  1. Physiotherapy Modalities (Preparation):
     Hot Pack Therapy: Applied to the lumbar region for 10-15 minutes before exercises to reduce muscle stiffness and pain.
     Interferential Therapy (IFT): Applied to the lower back for 10-15 minutes to decrease pain and improve circulation.
  2. Exercise Program (30-40 minutes per session, 3 times/week):
  A. Lumbar Stabilization Exercises
  B. Core Strengthening Exercises:
  Interventions: Other: Exercises for lower back
- Group receive Exercise and Physical Activity program (Experimental)
  Interventions: Other: Exercises and Physical Activity Program
- control (Other): control group (advices)
  Interventions: Other: Advices

INTERVENTIONS:
Other: Exercises for lower back — 1. Physiotherapy Modalities (Preparation):
     Hot Pack Therapy: Applied to the lumbar region for 10-15 minutes before exercises to reduce muscle stiffness and pain.
     Interferential Therapy (IFT): Applied to the lower back for 10-15 minutes to decrease pain and improve circulation.
  2. Exercise Program (30-40 minutes per session, 3 times/week):
  A. Lumbar Stabilization Exercises:
  B. Core Strengthening Exercises:
  Arms: Group receive Exercises
Other: Exercises and Physical Activity Program — 1. Frequency & Duration:
     Frequency: 3 days per week
     Duration: 30 to 40minutes per session
     Intensity: Low to moderate (RPE 11-13 on Borg scale; "light to somewhat hard")
  2. Warm-Up (5 minutes):
     Gentle walking on treadmill at slow speed (1.5-2.5 km/h)
     Light dynamic stretches for lower back, hips, and legs
  3. Main Activity
     A. Treadmill Walking:
     Speed: Comfortable pace for walking without pain
     Incline: Start flat, increase slightly (1-2%) if tolerated
     Goal: Promote cardiovascular endurance and safe weight-bearing activity
     B. Stationary Bicycle:
     Duration: 10-15 minutes
     Resistance: Low to moderate (enough to feel effort but no pain)
  4. Cool-Down (5 minutes):
     Slow treadmill walking or easy pedaling on the bike
     Gentle stretches: hamstrings, hip flexors, lumbar rotation
  5. Progression:
  based on patient tolerance Gradually in
  Arms: Group receive Exercise and Physical Activity program
Other: Advices — Advices
  Arms: control

SUMMARY:
This study evaluated the effects of a combined physical activity and structured exercise program on disability and mental health in elderly individuals suffering from chronic low back pain. Chronic low back pain is highly prevalent among older adults and is often associated not only with functional limitations and disability but also with psychological issues such as anxiety, depression, and poor sleep quality. Addressing both physical and mental health aspects is essential to improve overall well-being and quality of life in this population.

Participants in the study will be randomly assigned to one of three groups. The Exercise + Physical Activity Program Group received a structured exercise regimen specifically designed to improve core strength, flexibility, balance, and overall mobility. In addition to the exercise sessions, participants were provided with a tailored physical activity program aimed at promoting daily movement, reducing sedentary behavior, and enhancing functional capacity in their everyday life.

The Exercise-Only Group followed the same structured exercise regimen but did not receive the additional physical activity component, allowing for comparison of the effects of exercise alone versus combined interventions.

The Control Group continued with usual care, which included standard advice for managing low back pain but no structured exercise or physical activity intervention, serving as a baseline to evaluate the effectiveness of the other interventions.

Outcomes were assessed in terms of disability levels, measured using validated scales, as well as mental health parameters, including symptoms of depression, anxiety, and sleep quality. Post-intervention results indicated that participants in the combined exercise and physical activity group experienced the most significant improvements in functional ability, as reflected by reduced disability scores. This group also showed the largest reductions in symptoms of anxiety and depression and improvements in sleep quality. The exercise-only group demonstrated moderate improvements, highlighting the benefits of structured exercise alone, while the control group showed minimal changes in either physical function or mental health outcomes.

Measurements will be taken pre , post (8 weeks of PT interventions) and 8 weeks follow up

These findings emphasize the added value of integrating general physical activity into structured exercise programs. Incorporating daily movement and functional activity beyond formal exercise sessions appears to enhance both physical and psychological outcomes in elderly individuals with chronic low back pain. The study underscores the importance of a comprehensive approach in the management of chronic musculoskeletal pain in older adults, combining targeted exercise with strategies to increase overall daily activity levels.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 60 years or older.
2. Chronic Low Back Pain: History of low back pain lasting ≥12 weeks Poor sleep quality, defined as a Pittsburgh Sleep Quality Index (PSQI) score >5.
3. Mild to moderate symptoms of anxiety or depression, defined as a Hospital Anxiety and Depression Scale (HADS) score >7.
4. Ability to walk independently or with minimal assistance, allowing participation in treadmill or cycling exercises.

Exclusion Criteria:

1. Severe Mental Health Issues: Severe anxiety or depression (HADS score >15) or any other major psychiatric disorder.
2. Acute or Unstable Medical Conditions: Including recent cardiovascular events (e.g., myocardial infarction, unstable angina), uncontrolled hypertension, or severe respiratory disease.
3. Severe Musculoskeletal Disorders: Conditions that prevent safe participation in exercise, such as recent fractures, severe osteoporosis with risk of fracture, or advanced spinal pathology.
4. Neurological Disorders: Significant neurological impairments affecting balance or mobility (e.g., stroke, Parkinson's disease, severe peripheral neuropathy).
5. Recent Spine Surgery: Lumbar or spinal surgery within the past 6 months.
6. Cognitive Impairment: Inability to understand instructions or provide informed consent.
7. Participation in structured exercise programs in the past 3 months that could confound results.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
mental health | pre, 8 weeks post physiotherapy sessions and 8 weeks follow up
  Hospital Anxiety and Depression Scale (HADS) Symptoms of anxiety and depression were evaluated using the Hospital Anxiety and Depression Scale (HADS), a reliable and widely used instrument for assessing psychological distress in clinical and community populations. The HADS consists of 14 items, with 7 items measuring anxiety (HADS-A) and 7 measuring depression (HADS-D). Each item is scored from 0 to 3, resulting in subscale scores ranging from 0 to 21, with higher scores indicating more severe symptoms. The HADS is particularly suitable for elderly populations because it focuses on psychological symptoms rather than somatic complaints that could overlap with chronic physical conditions. In this study, changes in HADS scores provided insight into the impact of the interventions on mental health, helping to determine whether combining physical activity with structured exercises could alleviate anxiety and depressive symptoms associated with chronic low back pain.
Disability | pre, 8 weeks of physiotherapy session's and 8 weeks follow up
  Oswestry Disability Index (ODI) Functional disability related to chronic low back pain was measured using the Oswestry Disability Index (ODI), a validated questionnaire that assesses the impact of back pain on daily activities and overall functional ability. The ODI includes 10 sections covering pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and employment/homemaking. Each section is scored from 0 to 5, with the total score expressed as a percentage, where higher percentages indicate greater disability. The ODI is widely recognized as a gold standard for evaluating the severity of functional impairment in individuals with low back pain. In the present study, reductions in ODI scores following the interventions were used to quantify improvements in participants' physical function and independence, reflecting the effectiveness of both the structured exercise program and the additional physical activity regimen.
Sleep quality | pre Physiotherapy interventions, 8 weeks post and 8 follow up
  Pittsburgh Sleep Quality Index (PSQI) Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI), a widely validated self-report questionnaire designed to measure sleep disturbances and overall sleep quality over the past month. The PSQI evaluates seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored from 0 to 3, with higher scores indicating poorer sleep quality, and the global score ranges from 0 to 21. In this study, the PSQI was used to examine changes in sleep patterns and disturbances in elderly participants with chronic low back pain. Improvements in sleep quality were expected to reflect the effectiveness of the intervention in reducing pain-related sleep disruptions and enhancing overall mental and physical well-being.

IPD SHARING:
Plan to Share IPD: No